CLINICAL TRIAL: NCT05527054
Title: Analysis of Risk Factors of Diuretics Related Acute Kidney Injury in Hospitalized Patients and Development of Machine Learning Model
Brief Title: Risk Factors and Machine Learning Model for Diuretics Related Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xiao Li，MD, MD, Qianfoshan Hospital
Other Study IDs: LCYY-LX-20220101
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-11

CONDITIONS: Diuretic Toxicity; Acute Kidney Injury
Keywords: Diuretics; Aute kidney injury; Pharmacoepidemiology; Miss diagnosis; Risk factors; Logic regression
MeSH Terms: conditions — Acute Kidney Injury | interventions — Diuretics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI Group
  Interventions: Other: Diuretics
- Non-AKI Group
  Interventions: Other: Diuretics

INTERVENTIONS:
Other: Diuretics — Inpatients using diuretics

SUMMARY:
Acute kidney injury (AKI) is a series of clinical syndromes in which serum creatinine (Scr) concentrations increase over a short period of time, or urine output decreases. It has become an increasing global concern.Drug-induced acute kidney injury (D-AKI) refers to kidney injury caused by drugs or their metabolites within 7 days after the use of one or more drugs. The kidneys are rich in blood flow and have the function of acidifying the urine, making them an easy target for drug toxicity. Besides, there are enzymes in the kidney that metabolize some drugs, and if these drugs are metabolized abnormally in the kidney, substances toxic to the kidney may be produced.It was found that about 20% of AKI in hospitalized patients was caused by medications.Diuretics are one of the well-known nephrotoxic drugs, since they can directly or indirectly cause a significant decrease in renal blood perfusion and glomerular filtration rate through the mechanism of affecting tubulobulb feedback, which leads to kidney ischemia and hypoxia.However, there are few real-world studies on the incidence of AKI in hospitalized patients received diuretics. In this study, we aimed to explore the incidence and risk factors analysis of AKI in hospitalized patients received diuretics and develop the machine learning model for diuretics related AKI based on electronic medical record data. With the individual characteristics of patients, the risk of AKI can be evaluated before receiving diuretics, which may provide useful information for clinical decision making to better prevent D-AKI.

ELIGIBILITY:
Inclusion Criteria:

All inpatients who used diuretics during hospitalization Hospital stay ≥ 48h Age ≥ 18 years There were two or more blood creatinine tests during hospitalization

Exclusion Criteria:

Hospital stay < 48h Age < 18 years GFR < 30ml/min/1.73m2 within 48 hours after admission AKI was diagnosed on admission Less than two Scr test results during hospitalization The Scr values were always lower than 40 μmol/L during hospitalization Cases with incomplete medical history information

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were included if received treatment with diuretics and discharged from the hospital between January 1, 2018 and December 31, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | Through study completion，up to half a year.
  During the patient's hospitalization, acute kidney injury occurred after diuretic use.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao Li，MD, Jinan, Shandong, China